CLINICAL TRIAL: NCT06521216
Title: Comparing Different Oral Iron Dosing Regimens in Treatment of Iron Deficiency Anemia in Patients With Chronic Kidney Disease
Brief Title: Different Oral Iron Dosing Regimens in Treatment of Iron Deficency Anemia in Patients With Chronic Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Farrag Sayed Mohamed, Clinical physician, Assiut University
Other Study IDs: Oral iron in CKD patients
Record Dates: First submitted 2024-06-01; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: CKD
MeSH Terms: interventions — ferrous sulfate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients will receive oral iron in alternate day regimen: 50 patients will receive oral ferrous sulphate in alternate day regimen
  Interventions: Drug: Ferrous sulfate
- patients will receive oral iron in single daily dose regimen: 50 patients will receive oral ferrous sulphate in single daily dose regimen
  Interventions: Drug: Ferrous sulfate
- patients will receive oral iron in thrice daily dose regimen: 50 patients will receive oral ferrous sulphate in thrice daily dose regimen
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Ferrous sulfate — all patients will receive 200 mg elemental iron (ferrous sulphate)

SUMMARY:
Comparing between the efficacy of alternate day oral iron dose, once daily and thrice daily dose in improving anemia in CKD patients

DETAILED DESCRIPTION:
Anemia is common in chronic kidney disease (CKD) and has been associated with impaired quality of life, cardiovascular disease (CVD) and mortality.

Iron deficiency is common in patients with CKD and an important modifiable factor in treatment of anemia.

In particular, the Kidney Disease: Improving Global Outcomes (KDIGO) anemia work group guidelines define anemia in CKD as a hemoglobin concentration of <13.0 g/dL in men and <12.0 g/dL in women. The current guidelines recommend trial of iron supplementation in CKD when increase in hemoglobin concentration or decrease in erythropoietin dose is desired and investigations reveal percentage transferrin saturation (%TSAT) ≤ 30% and serum ferritin ≤ 500 ng/ml.

The absorption of iron from gastro-intestinal tract and release of iron from reticuloendothelial cells for erythropoiesis are tightly regulated through hepcidin-ferroportin axis. Hepcidin concentrations increase in response to iron excess and inflammation. CKD is associated with elevated hepcidin and ferritin concentrations due to underlying inflammation, independent of iron status.

Iron-deficiency anemia in individuals with CKD may result from functional iron deficiency, absolute iron deficiency, or both. The factors contributing to functional iron deficiency are chronic inflammation and poor hepcidin clearance seen in CKD, whereas absolute iron deficiency includes poor gastrointestinal (GI) dietary iron absorption and blood loss.

In patients with CKD who are not on dialysis, oral route may be preferred as initial mode of iron supplementation. Oral iron is inexpensive, self-administered, convenient and easily available.

Three different oral iron supplement strategies-once daily, multidose per day, and alternate-day dose-improve hemoglobin (Hgb) and iron indices in patients with iron deficiency anemia and chronic kidney disease (CKD).

Study showed that daily doses of oral iron reduced its absorption by increasing serum hepcidin levels. This study also found that administration of oral iron on alternate days as single doses improved iron absorption.

Theoretically, using lower doses and increasing time interval between consecutive doses might reduce the amount of unabsorbed iron in the gastrointestinal tract resulting in lesser gastrointestinal side effects. However, the major concern with alternate day dosing is that only half the total amount of iron is supplemented per unit time compared to daily dosing.

More recent data suggest that lower doses and infrequent administration may be as effective as the traditional regimen while probably associated with lower rates of adverse effects.

Investigators will investigate the effect of every other day, once daily and three times a day dosing of oral iron formulation on measures of iron sufficiency in patients with stages 2,3 and 4 CKD through a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients above 18 years old with CKD stages 2,3 and 4

Exclusion Criteria:

* CKD stage 5 (eGFR below 15 ).
* Patients with hemolytic anemias.
* Chronic liver diseases .
* Autoimmune diseases.
* Malignancy
* History of blood transfusion last 3 months before the study
* Pregnancy
* Adult polycystic kidney disease ( APCKD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients above 18 years old with CKD stages 2,3 and 4
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin level by gm/dl | 6 months
  Follow up Hemoglobin level in 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Farrag S Mohamed, Study Chair — Assiut University

REFERENCES:
- [Background] Stoffel NU, Cercamondi CI, Brittenham G, Zeder C, Geurts-Moespot AJ, Swinkels DW, Moretti D, Zimmermann MB. Iron absorption from oral iron supplements given on consecutive versus alternate days and as single morning doses versus twice-daily split dosing in iron-depleted women: two open-label, randomised controlled trials. Lancet Haematol. 2017 Nov;4(11):e524-e533. doi: 10.1016/S2352-3026(17)30182-5. Epub 2017 Oct 9. PMID 29032957
- See also: Sood, V., Kamboj, K., Bhatia, P. et al. A randomized trial of once daily versus twice daily dosing of oral iron in CKD. Sci Rep 13, 141 (2023). https://doi.org/10.1038/s41598-022-26589-x — https://rdcu.be/dJFpz